CLINICAL TRIAL: NCT06158178
Title: Evaluation of the Predictive Role of Choline PET/CT on the Survival of Patients Affected by Prostate Cancer.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PETCT-Chol-Survival
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic accuracy — The PET CT study with choline, being part of the normal standard diagnostic work-up of the patients, was performed following the normal clinical protocol. By analyzing the data retrospectively, the time elapsed following the prostatectomy operation and the follow up time after the choline PETCT study will be evaluated.

SUMMARY:
the increase in the serum PSA (prostate specific antigen) value following radical treatment commonly involves subsequent treatment which, in the absence of morphological evidence of disease recovery, is conducted empirically through local radiotherapy or systemic hormonal therapy. The use of PET with choline is therefore of extreme clinical interest as it allows to identify the site of disease recurrence, thus being able to direct towards a specific therapeutic treatment. The diagnostic accuracy of choline PET in identifying the location of the disease has been widely demonstrated in the literature and is comparable to those of conventional diagnostic methods previously described for the restaging of patients with prostatic disease. The real advantage of this method is the possibility of obtaining the same information as conventional methods by carrying out a single exam.

ELIGIBILITY:
Inclusion Criteria:

* adult patients suffering from prostate cancer who have undergone choline PET/TC

Exclusion Criteria:

* patients < 18 years

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: adult patients suffering from prostate cancer undergoing choline PET/CT at the San Raffaele hospital for restaging of the disease.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Choline PET-CT for the restaging of patients with prostatic disease. | 1 year
  By analyzing the data retrospectively, the time elapsed following the prostatectomy operation and the follow up time after the choline PETCT study will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No